CLINICAL TRIAL: NCT06806579
Title: Atezolizumab-bevacizumab and Other Immunotherapies: Real-life Experience for Treatment of Hepatocellular Carcinoma
Acronym: ARTE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ARTE
Record Dates: First submitted 2025-01-10; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: atezolizumab; bevacizumab; tremelimumab; durvalumab; immunotherapy; real-life; outcome
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
- Background Hepatocellular carcinoma (HCC), is the fifth most common cancer worldwide and the third leading cause of cancer-related death. In most cases (about 80%), HCC develops in a cirrhotic liver - a condition where the liver has been damaged over time, leading to scarring. This makes treatment more challenging.

This study will gather and analyze data from patients treated in real-world settings to:

1. Understand the effectiveness and safety of new treatment combinations (e.g., atezolizumab-bevacizumab and durvalumab-tremelimumab).

   Identify the best treatment sequences for patients with advanced liver cancer.
2. Discover clinical and laboratory markers that predict treatment responses, helping personalize care and optimize outcomes.

By addressing these questions, this study will provide valuable information to healthcare providers and guide future treatment decisions for patients with liver cancer.

DETAILED DESCRIPTION:
* Background Hepatocellular carcinoma (HCC), is the fifth most common cancer worldwide and the third leading cause of cancer-related death. In most cases (about 80%), HCC develops in a cirrhotic liver - a condition where the liver has been damaged over time, leading to scarring. This makes treatment more challenging.
* New Advances in Treatment Options

For many years, sorafenib was the only approved drug for advanced liver cancer when local treatments like surgery were not possible. However, significant advancements have changed the treatment landscape:

1. Atezolizumab and Bevacizumab (Immunotherapy Combination):

   In 2019, a groundbreaking study (ImBRAVE-150, Phase 3) demonstrated that combining atezolizumab (an immunotherapy drug) and bevacizumab (an anti-angiogenic drug) significantly improved disease-free survival (time without cancer worsening) and overall survival compared to sorafenib.

   This combination was approved in 2019 by the European Medicines Agency (EMA) and later by the Italian Medicines Agency (AIFA) in 2022.
2. Durvalumab and Tremelimumab (Dual Immunotherapy):

In February 2024, another combination-durvalumab and tremelimumab-was introduced following the results of the Phase 3 HIMALAYA trial, which also showed improved outcomes compared to sorafenib.

Several other immunotherapy-based combinations, such as camrelizumab-rivoceranib and nivolumab-ipilimumab, are under evaluation and may become available in the future.

* Why Is This Study Important?

  1. Real-World Effectiveness of Treatments:

     While clinical trials have shown promising results for atezolizumab-bevacizumab and durvalumab-tremelimumab, real-world data-information gathered from everyday clinical practice-are still limited. In particular, there is a lack of real-world evidence for the new durvalumab-tremelimumab combination. This study aims to fill that gap by collecting and analyzing data from patients treated in daily clinical practice.
  2. Understanding Treatment Sequences:

     After completing atezolizumab-bevacizumab or durvalumab-tremelimumab, what is the best next treatment? Currently, the only approved next-line drug is sorafenib, and for third-line treatment in Italy, cabozantinib is the only option. However, there is no clear scientific data on the effectiveness of these treatment sequences.

     As more therapies become available, it will be critical to identify the best sequence of treatments to extend survival and improve quality of life.
  3. Identifying Predictors of Response:

     Some patients respond better to treatment than others. This study seeks to identify clinical and laboratory markers that predict which patients will benefit most from specific therapies.

     For example, with sorafenib, the development of certain side effects (like skin reactions) was associated with better survival. It remains unclear whether similar markers exist for newer drug combinations.

     Additionally, the study will examine how factors such as treatment intolerance, patterns of disease progression, and second-line therapies influence survival outcomes.
* What This Study Aims to Achieve

This study will gather and analyze data from patients treated in real-world settings to:

1. Understand the effectiveness and safety of new treatment combinations (e.g., atezolizumab-bevacizumab and durvalumab-tremelimumab).

   Identify the best treatment sequences for patients with advanced liver cancer.
2. Discover clinical and laboratory markers that predict treatment responses, helping personalize care and optimize outcomes.

By addressing these questions, this study will provide valuable information to healthcare providers and guide future treatment decisions for patients with liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma not amenable to locoregional procedures
* Candidate to frontline systemic treatment with atezolizumab-bevacizumab or other immunotherapies

Exclusion Criteria:

* Concurrent treatment with other antineoplastic agents
* Other active neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from patients with hepatocellular carcinoma (HCC) who are candidates for treatment with atezolizumab-bevacizumab or durvalumab-tremelimumab. Patients will be evaluated in outpatient clinics or inpatient departments of the participating centers as part of the standard care pathway for HCC patients. Data will be collected at the patient's first evaluation and during subsequent assessments (approximately every 3-4 weeks), as per the routine care process for HCC patients receiving pharmacological treatments. The follow-up observation for each patient will continue as part of the standard care pathway.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate toxicity as first-line therapy | from enrollment up to 3 years from the first dose
  To evaluate toxicity of therapeutic sequences in which atezolizumab-bevacizumab or other immunothrapies were administered as first-line therapy within the standard care pathway for patients with hepatocellular carcinoma.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Progression-free survival | from enrollment up to 3 years from the first dose
  defined as the time between the first administration of atezolizumab-bevacizumab or durvalumab-tremelimumab and radiological progression
Overall survival | from enrollment up to 3 years from the first dose
  defined as the time between the treatment start and the death of the patient, or to the last follow-up evaluation
Objective response rate (ORR) | from enrollment up to 3 years from the first dose
  defined as the percentage of patients who achieve a partial or complete response to the disease on follow-up imaging, according to RECIST 1.1 criteria, out of the total number of patients who undergo at least one radiological assessment.
Rate of Patients Eligible for Second-Line Treatments | from enrollment up to 3 years from the first dose
  defined as the percentage of patients who, after the definitive discontinuation of atezolizumab-bevacizumab or other immunotherapies, have sufficiently good general conditions and liver function to allow the prescription of an additional line of systemic treatment.
Safety monitoring | from enrollment up to 3 years from the first dose
  Incidence of Adverse Events Related to Atezolizumab-Bevacizumab or other immunotherapies

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Tovoli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (24):
- Italy (24):
  - Ospedali Riuniti Ancona, Via Conca, 71, 60126 Torrette AN, Torrette, AN
  - I.R.C.C.S. "S. De Bellis", Via Turi, 27, 70013 Castellana Grotte BA, Castellana Grotte, BA
  - AUSL Bologna Via Castiglione 15 40136 Bologna BO, Bologna, BO
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna (Oncology Unit), Bologna, BO 40136, Bologna, BO
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna (Semiotics Unit), Bologna, BO
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione "Garibaldi, Piazza Santa Maria di Gesù, 5, 95123 Catania CT, Catania, CT
  - Ospedali Riuniti. Viale Pinto Luigi, 1, 71122 Foggia FG., Foggia, FG
  - Ospedali Riuniti. Viale Pinto Luigi, 1, 71122 Foggia FG, Foggia, FG
  - AOU Careggi. Largo G. Alessandro Brambilla, 3. 50134 Firenze FI, Florence, FI
  - Policlinico di Modena Via del Pozzo, 71, 41125 Modena MO, Modena, Missouri
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico. via Francesco Sforza, 28 - 20122 Milano., Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Piazza dell'Ospedale Maggiore, 3, 20162 Milano, Milan, MI
  - Humanitas Research Hospital. Via Alessandro Manzoni, 56, 20089 Rozzano MI, Rozzano, MI
  - Azienda Ospedaliero- Universitaria Paolo Giaccone. Via Liborio Giuffrè, 5, 90127 Palermo, Palermo, PA
  - Istituto Oncologico Veneto. Via Gattamelata, 64, 35128 Padova PD, Padua, PD
  - AOU Pisana. Via Roma 67. 56126 Pisa PI, Pisa, PI
  - Ospedale degli Infermi Viale Stradone, 9 48018 Faenza (RA), Faenza, RA
  - IRCCS Santa Maria Nuova Viale Risorgimento, 80, 42123 Reggio Emilia, Reggio Emilia, RE
  - Policlinico Gemelli. Largo Agostino Gemelli, 8, 00168 Roma RM, Roma, RM
  - Azienda sanitaria universitaria Friuli Centrale, Piazzale Santa Maria della Misericordia, 15 33100 Udine (UD), Udine, UD
  - Azienda Ospedaliera Universitaria Integrata di Verona. Piazzale Aristide Stefani, 1, 37126 Verona VR, Verona, VR
  - P.O. Ospedale del Mare. Via Enrico Russo, 11, 80147 Napoli NA, Napoli
  - Azienda Ospedaliero- Universitaria Maggiore della Carità, Padiglione G, L.go Bellini, 28100 Novara NO, Novara

IPD SHARING:
Plan to Share IPD: Undecided
Privacy regulations

REFERENCES:
- See also: link to full text paper (open access) — https://pubmed.ncbi.nlm.nih.gov/39168753/